CLINICAL TRIAL: NCT03398785
Title: An Open-label, Prospective, Controlled Clinical Trial on Effects and Safety of Adrenal Artery Ablation (Triple A) for Primary Aldosteronism
Brief Title: Adrenal Artery Ablation Treats Primary Aldosteronism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Triple A-PA
Record Dates: First submitted 2017-12-24; First posted 2018-01-12 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Primary Aldosteronism; Hypertension
Keywords: Primary Aldosteronism; Hypertension; Ablation; Adrenal Gland
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Intervention Model Description: Patients in the Intervention group will be treated with endovascular chemical ablation of adrenal gland by endovascular injection of dehydrated alcohol. Patients in the Control group will be treated with conventional anti-hypertensive drugs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intevention (Experimental): Adrenal Artery Ablation
  Interventions: Procedure: Endovascular chemical Ablation of Adrenal Gland
- Control (No Intervention): No intervention, but treated with standard anti-hypertensive drigs

INTERVENTIONS:
Procedure: Endovascular chemical Ablation of Adrenal Gland — Patients in this group will be treated with partial ablation of adrenal gland by endovascular injection of dehydrated alcohol.
  Arms: Intevention

SUMMARY:
Primary aldosteronism (PA) is one of the most common cause of endocrine and resistant hypertension. Current studies have shown that the activation of the renin-angiotensin-aldosterone system (RAAS) and the increased sympathetic nerve activity in the central or local tissue are the key mechanisms of high blood pressure and its organ damages.

The classical method for diagnosis of primary aldosteronism depends on the detection of peripheral venous blood aldosterone level, which is incapable of accurate positioning diagnosis. On the other hand, the current guidelines recommend that surgery and aldosterone receptor inhibitors were the only treatment for primary aldosteronism. However, only about 35% of aldosterone tumors and a small part of unilateral adrenal hyperplasia can be treated by surgery. More than 60% of idiopathic aldosteronism and bilateral adrenal hyperplasia need long-term drug therapy. However, long-term aldosterone inhibitor treatment may also cause hyperkalemia, male breast hyperplasia, female hirsutism and other adverse reactions.

Therefore, the investigators proposed that endovascular chemical partial ablation of the adrenal gland can lower the aldosterone level, reduce the blood pressure and recover the potassium metabolism balance. In order to confirm the above effects, the investigators conduct an open, prospective, positive controlled study in patients with primary aldosteronism patients (including aldosterone, idiopathic aldosteronism and adrenal hyperplasia). The effects on blood pressure, blood electrolytes, adrenal hormones, metabolic indexes, target organ damages were observed to explore the efficacy and safety of the endovascular ablation of the adrenal gland in the treatment of primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Primary Aldosteronis diagnosed by increased Renin ratio (ARR) and serum aldosterone levels ≥15 ng / dl, and confirmed by saline injection test or captopril inhibition test.
* Idiopathic aldosteronism, bilateral adrenal hyperplasia, and unilateral adrenal hyperplasia with no superior secretion confirmed with adrenal CT and adrenal venous blood (AVS).
* The patients was diagnosed with aldosteronoma or unilateral adrenal hyperplasia but refused to surgical excision.
* Signed informed consent and agreed to participate in this study.

Exclusion Criteria:

* Aldosterone cancer.
* Hyperkalemia.
* Renal failure or the following history of nephropathy: serum creatinine 1.5 times higher than the upper limit; dialysis history; or nephrotic syndrome.
* Secondary hypertension except the primary aldosteronism.
* Adrenergic insufficiency.
* Heart failure with NYHA grade Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders, drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 2 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Any surgical or medical condition which can significantly alter the absorption, distribution, metabolism, or excretion of any study drug.
* Allergy or any contraindications for the study drugs, contrast agents and alcohol.
* Refused to sign informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change of 24-h average systolic blood pressure compared with the baseline | 24 weeks
  Change of 24-h average systolic blood pressure compared with the baseline at the end of the study (24 weeks) in the intervention group.

SECONDARY OUTCOMES:
Change of 24-h average systolic blood pressure between two groups | 24 weeks
  Change of 24-h average systolic blood pressure between the intervention and control group at the end of the study (24 weeks)
Change of anti-hypertensive regimen between two groups | 24 weeks
  Change of number, classes, and combinations of classes of antihypertensive drugs between the intervention and control group at the end of the study (24 weeks)
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between two groups | 24 weeks
  Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group at the end of the study (24 weeks)
Change of office systolic and diastolic pressure between two groups | 24 weeks
  Change of office systolic and diastolic pressure between the intervention and control group at the end of the study (24 weeks)
Change of blood electrolytes（serum potassium and natrium in mmol/L） | 24 weeks
  Change of blood electrolytes（serum potassium and natrium in mmol/L） compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of plasma aldosterone and 24-h urine aldosterone | 24 weeks
  Change of plasma aldosterone and 24-h urine aldosterone compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of plasma renin | 24 weeks
  Change of plasma renin compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of plasma cortisol and 24-h urine cortisol | 24 weeks
  Change of plasma cortisol and 24-h urine cortisol compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of liver enzymes (ALT, AST) | 24 weeks
  Change of liver enzymes (ALT, AST) compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of serum creatinine | 24 weeks
  Change of serum creatinine compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of fasting blood glucose | 24 weeks
  Change of fasting blood glucose in mmol/L compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L | 24 weeks
  Change of lipids profiles (Total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglyceride) in mmol/L compared with baseline, and between the intervention and control group at the end of the study (24 weeks)

OTHER OUTCOMES:
Change of testosterone and estrogen levels | 24 weeks
  Change of testosterone and estrogen levels compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of 24-h urine microalbumin, microalbumin/creatinine ratio | 24 weeks
  Change of 24-h urine microalbumin, microalbumin/creatinine ratio compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, LVEF, LVM) | 24 weeks
  Change of parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, LVEF, LVM) compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of carotid intima-media thickness assessed by carotid ultrasound | 24 weeks
  Change of carotid intima-media thickness(CIMT) assessed by carotid ultrasound compared with baseline, and between the intervention and control group at the end of the study (24 weeks)
Change of electrocardiogram manifestations | 24 weeks
  Change of electrocardiogram manifestations(heart rhythms, heart rates and arrhythmia ) compared with baseline, and between the intervention and control group at the end of the study (24 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun F, Hong Y, Zhang H, Liu X, Zhao Z, He H, Yan Z, Zhu Z. Determination of adrenal hypersecretion in primary Aldosteronism without aldosterone-production adenomas. BMC Endocr Disord. 2021 May 31;21(1):114. doi: 10.1186/s12902-021-00770-1. PMID 34059026